CLINICAL TRIAL: NCT04893460
Title: A Mobile App Based Cognitive Dissonance Intervention for Smoking Cessation
Brief Title: CoQuit Study for Smoking Cessation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Research Behavioral Intervention Strategies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DP006495-01
Record Dates: First submitted 2021-05-14; First posted 2021-05-19 (Actual); Results first posted 2025-09-04 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): All participants will use the CoQuit App for Smoking Cessation
  Interventions: Behavioral: CoQuit App

INTERVENTIONS:
Behavioral: CoQuit App — The CoQuit App is a cognitive dissonance based app for smoking cessation.

SUMMARY:
This study investigated the feasibility of a cognitive dissonance-based mobile app for smoking cessation (CDI). Cognitive dissonance refers to the conflict between beliefs and behaviors; interventions are designed to promote this conflict to motivate people to change their behavior. Recent research has demonstrated the efficacy and potential of using cognitive dissonance interventions for a wide range of health and behavioral problems including smoking cessation. This study developed an initial version of the CDI mobile app and evaluated the app in an evaluation study with 60 adult smokers.

DETAILED DESCRIPTION:
An initial version of the CoQuit app was developed and tested with 60 adult smokers. All participants were recruited through social media and were screened and consented online. After enrolling, participants received a link to the baseline survey which asked about past and current tobacco use, nicotine dependence, motivation to quit, cognitive dissonance and demographic information. All participants were assigned to an online support group of 5 or 6 people. The group received simultaneous invites to the app so they were able to move through the 25 day program together. The app contained short videos of a CoQuit facilitator who presented instructions for specific tasks, such as writing a brief letter to a friend or family member explaining their commitment to stop smoking. Participants recorded videos of themselves related to these activities and posted the videos within the app where they were viewed by other members of the group. All participants completed a six weeks post baseline online assessment asking about past and current tobacco use, quit attempts, as well as feedback on usability and possible improvements to the app.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Self-reported daily smoking
* Having a valid home mailing address
* English speaking
* Access to a smart phone with video capability and internet
* Expressed desire to quit smoking

Exclusion Criteria:

* Currently participating in any tobacco cessation programs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-09-29 (Actual); Study Completion 2021-09-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dana Smith, PhD, Principal Investigator — Influents Innovations/Oregon Research Institute; Herb Severson, PhD, Principal Investigator — Influents Innovations/Oregon Research Institute
Locations (1):
- ORBIS/Oregon Research Institute, Springfield, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention
Started | 72
Completed | 54
Not Completed | 18
Not completed — Lost to Follow-up | 18

BASELINE CHARACTERISTICS:
Arm/Group | Intervention
Number analyzed (Participants) | 72
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.4 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55
  Male | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 59
  More than one race | 1
  Unknown or Not Reported | 7
Education Level [Count of Participants; unit: Participants]
  Did not graduate high school | 2
  High school graduate | 10
  Some college, no degree | 26
  Technical school or Associate degree | 16
  Bachelor degree | 11
  Master degree | 6
  Doctorate degree | 1

OUTCOME MEASURES:

1. Primary Outcome: Cognitive Dissonance
Description: Participants were asked to give a "gut-level response" to 14 words used to describe various attributes of cognitive dissonance (e.g., uncomfortable, shame). Response options for each attribute were on a 7-point scale (1 = does not apply at all, 7 = applies very much). A mean score was computed across all 14 words. A higher score was associated with greater levels of cognitive dissonance. In addition to the baseline and six-week follow-up assessment of cognitive dissonance, participants were asked five times during the 25 days of using the app. The five times were after completing the "Costs" activity on day 3, the "Quit Letter" activity on day 6, the "Planning for Pitfalls" activity on day 10, the "Staying Smoke Free" activity on day 14, and the "Letter to Youth" activity on day 19.
Time Frame: Baseline, 5 times during app use (days 3, 6, 10, 14 and 19 of the 25 day program), Six weeks post baseline
Population: Due to conceptual concerns about imputing smoking status, decreases in smoking from pretest to posttest were evaluated with participants who completed both the pretest and posttest assessment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 54
units on a scale
  Baseline | 2.23 (1.23)
  In app 1 - After Costs Activity | 3.32 (1.43)
  In app 2 - After Quit Letter Activity | 4.33 (1.48)
  In app 3 - After Pitfalls Activity | 3.67 (1.76)
  In app 4 - After Smoke Free Activity | 3.14 (1.83)
  In app 5 - After Letter to Youth Activity | 3.69 (1.89)
  6 Weeks Post Baseline | 2.48 (1.34)
Statistical Analysis 1: Comparison: Intervention; Test type: Superiority — This model is a paired t-test that tests for change in cognitive dissonance from baseline to after the Cost activity; p = .003, t-test, 2 sided; Mean Difference (Final Values) = -1.09, Standard Error of Mean 0.33
Statistical Analysis 2: Comparison: Intervention; This model is a paired t-test that tests for change in cognitive dissonance from baseline to after the Quit Letter activity; Test type: Superiority; p < .001, t-test, 2 sided; Mean Difference (Final Values) = -2.10, Standard Error of Mean 0.44
Statistical Analysis 3: Comparison: Intervention; This model is a paired t-test that tests for change in cognitive dissonance from baseline to after the Pitfalls activity; Test type: Superiority; p = .004, t-test, 2 sided; Mean Difference (Final Values) = -1.44, Standard Error of Mean 0.41
Statistical Analysis 4: Comparison: Intervention; This model is a paired t-test that tests for change in cognitive dissonance from baseline to after the Smoke Free activity; Test type: Superiority; p = .098, t-test, 2 sided; Mean Difference (Final Values) = -0.91, Standard Error of Mean 0.48
Statistical Analysis 5: Comparison: Intervention; This model is a paired t-test that tests for change in cognitive dissonance from baseline to after the Letter to Youth activity; Test type: Superiority; p = .042, t-test, 2 sided; Mean Difference (Final Values) = -1.46, Standard Error of Mean 0.68
Statistical Analysis 6: Comparison: Intervention; This model is a paired t-test that tests for change in cognitive dissonance from baseline to 6 weeks post baseline; Test type: Superiority; p = .364, t-test, 2 sided; Mean Difference (Final Values) = -0.25, Standard Error of Mean 0.22

2. Primary Outcome: Number of Participants With Number Cigarettes Smoked Per Day
Description: A one-item question that asked about the number of cigarettes smoked per day. Response options were on a 6-point scale, where 1 = 5 or less, 2 = 6-10, 3 = 11-15, 4 = 16-20, 5 = 21-30, and 6 = 31 or more. A higher score indicates a greater number of cigarettes smoked per day.
Time Frame: Baseline and Six Weeks Post Baseline
Population: Due to conceptual concerns about imputing smoking status, decreases in smoking from pretest to posttest was evaluated with participants who completed both the pretest and posttest number of cigarettes smoked item.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention
Number analyzed (Participants) | 46
Participants
  Baseline: 5 or less | 0
  Baseline: 6-10 | 12
  Baseline: 11-15 | 13
  Baseline: 16-20 | 10
  Baseline: 21-30 | 11
  Baseline: 31 or more | 0
  6 Weeks Post Baseline: 5 or less | 13
  6 Weeks Post Baseline: 6-10 | 16
  6 Weeks Post Baseline: 11-15 | 5
  6 Weeks Post Baseline: 16-20 | 9
  6 Weeks Post Baseline: 21-30 | 3
  6 Weeks Post Baseline: 31 or more | 0
Statistical Analysis 1: Comparison: Intervention; The non-parametric Wilcoxon signed-rank test was used to evaluate whether participants were smoking fewer cigarettes per day; Test type: Superiority; p < .001, Wilcoxson Signed Rank Test; median pairwise average = 17.67

3. Secondary Outcome: Readiness to Quit
Description: Participants were asked to rate what best describes how they currently think about quitting smoking. The one item had a 1-point scale (0 = I have no thought about quitting smoking, 2 = I think I need to consider quitting smoking someday, 5 = I think I should quit smoking, but I am not quite ready, 8 = I am starting to think about how to reduce the number of cigarettes I smoke a day, 10 = I am taking action to quit smoking, 11 = I have stopped smoking). A higher score was associated with greater readiness to quit smoking. In addition to the baseline and six-week follow-up assessment of readiness to quit, participants were asked five times during the 25 days of using the app. The five times were after completing the "Costs" activity on day 3, the "Quit Letter" activity on day 6, the "Planning for Pitfalls" activity on day 10, the "Staying Smoke Free" activity on day 14, and the "Letter to Youth" activity on day 19.
Time Frame: Baseline, 5 times during app use (days 3, 6, 10, 14 and 19 of the 25 day program), Six weeks post baseline
Population: Due to conceptual concerns about imputing smoking data, readiness to quit from was evaluated with participants who completed both the pretest and posttest readiness items.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 46
units on a scale
  Baseline | 7.52 (1.63)
  In app 1 - After Costs Activity | 7.64 (2.20)
  In app 2 - After Quit Latter Activity | 8.24 (1.81)
  In app 3 - After Pitfalls Activity | 8.81 (1.54)
  In app 4 - After Smoke Free Activity | 8.50 (1.86)
  In app 5 - After Letter to Youth Activity | 8.93 (1.75)
  6 week Post Baseline | 7.50 (2.08)
Statistical Analysis 1: Comparison: Intervention; Test type: Superiority — This model is a paired t-test that tests for change in readiness to quit smoking from baseline to after the Cost activity; p = .776, t-test, 2 sided; Mean Difference (Net) = -0.12, Standard Error of Mean 0.42
Statistical Analysis 2: Comparison: Intervention; Test type: Superiority — This model is a paired t-test that tests for change in readiness to quit smoking from baseline to after the Quit Latter activity; p = .219, t-test, 2 sided; Mean Difference (Final Values) = -0.72, Standard Error of Mean 0.45
Statistical Analysis 3: Comparison: Intervention; Test type: Superiority — This model is a paired t-test that tests for change in readiness to quit smoking from baseline to after the Pitfalls activity; p = .043, t-test, 2 sided; Mean Difference (Final Values) = -1.29, Standard Error of Mean 0.55
Statistical Analysis 4: Comparison: Intervention; Test type: Superiority — This model is a paired t-test that tests for change in readiness to quit smoking from baseline to after the Smoke Free activity; p = .219, t-test, 2 sided; Mean Difference (Final Values) = -0.98, Standard Error of Mean 0.67
Statistical Analysis 5: Comparison: Intervention; Test type: Superiority — This model is a paired t-test that tests for change in readiness to quit smoking from baseline to after the Letter to Youth activity; p = .110, t-test, 2 sided; Mean Difference (Final Values) = -1.41, Standard Error of Mean 0.54
Statistical Analysis 6: Comparison: Intervention; Test type: Superiority — This model is a paired t-test that tests for change in readiness to quit smoking from baseline to 6 week post baseline assessment; p = .868, t-test, 2 sided; Mean Difference (Final Values) = 0.02, Standard Error of Mean 0.26

ADVERSE EVENTS:
Time Frame: 6 weeks
Arm/Group | Intervention
All-Cause Mortality (participants affected / at risk) | 0/72
Serious Adverse Events (participants affected / at risk) | 0/72
Other Adverse Events (participants affected / at risk) | 0/72

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2020-05-05): https://cdn.clinicaltrials.gov/large-docs/60/NCT04893460/Prot_SAP_ICF_000.pdf